CLINICAL TRIAL: NCT00640991
Title: An International Multicentre Randomized Controlled Trial of Intensive Insulin Therapy Targeting Normoglycemia In Acute Myocardial Infarction: the RECREATE (REsearching Coronary REduction by Appropriately Targeting Euglycemia) Pilot Study
Brief Title: REsearching Coronary REduction by Appropriately Targeting Euglycemia (RECREATE Pilot Study)
Acronym: RECREATE Pilot
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Dr. Hertzel Gerstein, Professor of Medicine, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECREATE Pilot
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Hyperglycemia; Cardiovascular Diseases; Myocardial Infarction
Keywords: Clinical Trial; Insulin
MeSH Terms: conditions — Hyperglycemia; Cardiovascular Diseases; Myocardial Infarction; Insulin Resistance | interventions — insulin glulisine; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Patients assigned to the control arm will receive usual care for AMI, according to local practice of each participating centre.
- Intervention (Experimental): The experimental arm will have an IV infusion of glulisine insulin started directly after randomization for at least 24 hours and for as long as CCU-level care is required, and the insulin infusion will be adjusted to achieve and maintain a target glucose range of 5.0-6.6 mmol/L (90-118 mg/dL). Once transferred to the ward, patients in the experimental arm will switch to glargine insulin and will continue this treatment for the remainder of their hospitalization and after hospital discharge, for a total duration of 30 days post randomization.
  Interventions: Drug: glulisine insulin, glargine insulin

INTERVENTIONS:
Drug: glulisine insulin, glargine insulin — IV infusion of glulisine, SC injection of glargine
  Other Names: Apidra, Lantus
  Arms: Intervention

SUMMARY:
Insulin will safely reduce glucose levels in patients with acute ST-elevation myocardial infarction and admission hyperglycemia.

DETAILED DESCRIPTION:
Patients will be randomly assigned to either the control arm and will receive usual AMI care or the experimental arm, which will include routine AMI care as well as intensive therapy intervention.

In addition to the capillary blood glucose measurements obtained to titrate insulin doses in the experimental arm patients, laboratory plasma glucose will be drawn in all patients at randomization, 10, 24, 48, and 72 hours post randomization, 7 days post randomization (or hospital discharge if that occurs first), and 30 days post randomization.

ELIGIBILITY:
Inclusion Criteria:

Both nondiabetic patients and patients with non-insulin-requiring type 2 diabetes mellitus admitted with a suspected AMI are eligible if they meet the following criteria:

* Signs or symptoms of AMI with definite ECG changes, defined as persistent ST-segment elevation (> or = than 1 mm)in two or more contiguous leads, or new left bundle branch block
* Onset of symptoms within 24 hours before hospital presentation
* Capillary blood glucose level on presentation > or = 8.0 mmol/L (144 mg/dL)

Exclusion Criteria:

* Patient with conditions that REQUIRE the administration of insulin, including:

  * Type 1 diabetes mellitus, defined by a documented history of diabetes mellitus before the age of 30
  * Type 2 diabetes mellitus that was treated with insulin prior to AMI presentation
  * Type 2 diabetes mellitus that is known to be very poorly controlled (e.g. admission capillary blood glucose > 16.0 mmol/L (288 mg/dL)or marked elevation in glucose for which the site investigator plans to treat with insulin therapy)
* A history of severe hypoglycemic episodes (defined as hypoglycemia with symptoms which the patient is unable to reverse without the assistance of another person) within the past two years
* Known or suspected end-stage liver disease (due to the risk of hypoglycemia in the setting of liver dysfunction and consequent impaired regulation of glucose homeostasis)
* Cardiogenic shock on admission (due to the inaccuracy of glucose meter readings)
* Documented pregnancy
* Any concomitant disease (e.g. cancer) that might limit life expectancy to less than 90 days
* Anticipated poor adherence with study treatments or an other factor that might jeopardize 90-day follow-up (e.g. no fixed address, long distance to hospital, etc.)
* Prior enrollment in this trial or current enrollment in another trial of ST-segment elevation myocardial infarction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The 24-hour difference in mean glucose between the two study groups. | 24 hours

SECONDARY OUTCOMES:
The difference in mean glucose level achieved at 7 days or hospital discharge (whichever is first) | 7 days or discharge
The difference in mean glucose level achieved at 30 days between study groups | 30 days
Nonfatal recurrent myocardial infarction, nonfatal stroke, or cardiovascular death (as a composite and as separate outcomes) | Discharge, 30 days, 90 days, 1 year
Rehospitalization for congestive heart failure | Discharge, 30 days, 90 days, 1 year
All cause mortality | Discharge, 30 days, 90 days, 1 year
Resuscitated cardiac arrest or life-threatening arrhythmia (as a composite and as separate outcomes) | Discharge, 30 days, 90 days, 1 year
Cardiogenic shock | Discharge, 30 days, 90 days, 1 year
Cardiac procedures | Discharge, 30 days, 90 days, 1 year
Rehospitalization for any cause | Discharge, 30 days, 90 days, 1 year
Symptomatic and severe hypoglycemic episodes | Discharge, 30 days, 90 days, 1 year
Hypokalemic episodes | Discharge

CONTACTS AND LOCATIONS:
Overall Officials: Hertzel Gerstein, MD, MSc, FRCPC, Principal Investigator — McMaster University; Salim Yusuf, DPhil, FRCPC, FRSC, Principal Investigator — McMaster University
Locations (13):
- Instituto Medico Adrogue, Adrogué, Buenos Aires, Argentina
- Hamilton Health Sciences, General Site, Hamilton, Ontario, Canada
- India (11):
  - Assam Medical College Hospital, Dt. Dibrugarh, Assam
  - Lifeworth Super Specialty Hospital, Raipur, Chhattisgarh
  - Post Graduate Institute of Medical, Rohtak, Haryana
  - St. Johns Medical College, Bangalore, Karnataka
  - Nanjappa Hospital, Shimoga, Karnataka
  - Baby Memorial Hospital, Calicut, Kerala
  - Caritas Hospital, Kottayam, Kerala
  - KEM Hospital, Mumbai, Maharashtra
  - MGIMS, Wardha, Maharashtra
  - Railway Hospital, Chennai, Tamil Nadu
  - Avanti Institute of Cardiology, Nagpur